CLINICAL TRIAL: NCT04784260
Title: Microbiome Influence on Seminal Quality on Semen Donors
Brief Title: Microbiome Influence on Seminal Quality
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI Alicante (Other)
Responsible Party: Sponsor
Other Study IDs: 1911-ALC-100-ES
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-02

CONDITIONS: Infertility, Male
Keywords: Microbiome; Semen
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (normozoospermic): >15 mill/ml and >32% progressive mobility.: Analysis of the microbiome by extracting DNA from ejaculates, amplification of bacterial DNA with feeders aimed at the regions of the bacterial rRNA 16 S gene, sequencing, library preparation and bioinformatic analysis.
  Interventions: Other: Microbiome analysis
- Group B (normozoospérmic): <15 mill/ml and <32% progressive mobility.: Analysis of the microbiome by extracting DNA from ejaculates, amplification of bacterial DNA with feeders aimed at the regions of the bacterial rRNA 16 S gene, sequencing,library preparation and bioinformatic analysis.
  Interventions: Other: Microbiome analysis

INTERVENTIONS:
Other: Microbiome analysis — Evaluate the bacterial composition in sperm from the different groups

SUMMARY:
The microbiome plays an important role in health and in some unknown etiologies. Some previous studies have identified bacteria in semen as a potential factor in male infertility. More studies are needed to discover associations between microbiomes and semen quality. In this study, forty semen samples from donors candidates will be collected where clinical criteria for seminal quality (volume, concentration, motility and morphology) will be measured and bacterial communities examined. With the next-generation sequencing of gene technology and bioinformatic analysis, we can investigate the associations between bacterial communities and seminal quality. It would be interesting to know if the proportion of certain bacteria is significantly higher in samples of normal seminal quality or significantly higher in samples of low seminal quality. This study could contribute to the current understanding of certain etiologies of male fertility.

DETAILED DESCRIPTION:
Surplus semen samples will be collected from donor candidates who come to the IVI Alicante clinic with ages between 18 and 35 years old and who intend to participate in the donation program for the semen bank, and come to evaluate their quality. Informed consent for this study will be given to all of them, which they will have to return signed.

Depending on the semen quality evaluated in the diagnostic sample within the usual practice, in the laboratory the participants will be divided into 2 groups according to the WHO reference values in terms of sperm concentration and percentage of progressive motility:

* Group A (Normozoospermics): ≥15 mill / ml and> 32% progressive mobility.
* Group B (Non-normozoospermic): <15 mill / ml and <32% progressive mobility. The study will consist of 2 years. The first year will be used to collect all the diagnostic seminal samples from donor candidates, and the second year will be used in its first months to analyze the microbiome by extracting DNA from ejaculates, amplifying bacterial DNA with targeted primers. to the bacterial 16S rRNA gene regions, sequencing, library preparation and bioinformatic analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years. Suitable on your first informational visit.

Exclusion Criteria:

* Presence of own or hereditary pathology. Presence of mental or behavioral disturbance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include those donor candidates who come to undergo the diagnostic spermiogram within the usual practice and who have previously undergone an informative visit about the donation program and have been accepted for their profile and anamnesis regarding their family history and of health.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Seminal quality and microbiome | Two years
  Evaluate the bacterial composition of semen in a given population (sperm donor) analyzing the microbiome by extracting DNA from ejaculates, amplifying bacterial DNA with targeted primers to the bacterial 16S rRNA gene regions, sequencing, library preparation and bioinformatic analysis.

SECONDARY OUTCOMES:
Microbiome and individual semen quality parameters Microbiome as a fertility biomarker | seven months
  To assess whether the composition of the microbiome affects the different seminal quality parameters studied differently (concentration, mobility,...) It would be interesting with these findings to study the possibility of finding biomarkers that indicate that the presence of certain microorganisms may negatively or positively affect seminal quality and, that either by the presence or absence of these, they can help us to find a relationship with the seminal parameters studied, in order to find a cause and a possible treatment that can improve. In addition, see if it would help improve the diagnosis of infertility cases where there is no other apparent cause.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sellés, PhD, Principal Investigator — Instituto Valenciano de Infertilidad, IVI Alicante
Locations (1):
- IVI Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rittenberg V, El-Toukhy T. Medical treatment of male infertility. Hum Fertil (Camb). 2010 Dec;13(4):208-16. doi: 10.3109/14647273.2010.534833. PMID 21117930
- [Background] Weng SL, Chiu CM, Lin FM, Huang WC, Liang C, Yang T, Yang TL, Liu CY, Wu WY, Chang YA, Chang TH, Huang HD. Bacterial communities in semen from men of infertile couples: metagenomic sequencing reveals relationships of seminal microbiota to semen quality. PLoS One. 2014 Oct 23;9(10):e110152. doi: 10.1371/journal.pone.0110152. eCollection 2014. PMID 25340531
- [Background] Marchesi JR, Ravel J. The vocabulary of microbiome research: a proposal. Microbiome. 2015 Jul 30;3:31. doi: 10.1186/s40168-015-0094-5. eCollection 2015. PMID 26229597
- [Background] Altmae S, Franasiak JM, Mandar R. The seminal microbiome in health and disease. Nat Rev Urol. 2019 Dec;16(12):703-721. doi: 10.1038/s41585-019-0250-y. Epub 2019 Nov 15. PMID 31732723
- [Background] Cox MJ, Cookson WO, Moffatt MF. Sequencing the human microbiome in health and disease. Hum Mol Genet. 2013 Oct 15;22(R1):R88-94. doi: 10.1093/hmg/ddt398. Epub 2013 Aug 13. PMID 23943792
- [Background] Koedooder R, Mackens S, Budding A, Fares D, Blockeel C, Laven J, Schoenmakers S. Identification and evaluation of the microbiome in the female and male reproductive tracts. Hum Reprod Update. 2019 May 1;25(3):298-325. doi: 10.1093/humupd/dmy048. PMID 30938752
- [Background] Monteiro C, Marques PI, Cavadas B, Damiao I, Almeida V, Barros N, Barros A, Carvalho F, Gomes S, Seixas S. Characterization of microbiota in male infertility cases uncovers differences in seminal hyperviscosity and oligoasthenoteratozoospermia possibly correlated with increased prevalence of infectious bacteria. Am J Reprod Immunol. 2018 Jun;79(6):e12838. doi: 10.1111/aji.12838. Epub 2018 Mar 3. PMID 29500854
- [Background] Gevers D, Knight R, Petrosino JF, Huang K, McGuire AL, Birren BW, Nelson KE, White O, Methe BA, Huttenhower C. The Human Microbiome Project: a community resource for the healthy human microbiome. PLoS Biol. 2012;10(8):e1001377. doi: 10.1371/journal.pbio.1001377. Epub 2012 Aug 14. PMID 22904687
- [Background] Hou D, Zhou X, Zhong X, Settles ML, Herring J, Wang L, Abdo Z, Forney LJ, Xu C. Microbiota of the seminal fluid from healthy and infertile men. Fertil Steril. 2013 Nov;100(5):1261-9. doi: 10.1016/j.fertnstert.2013.07.1991. Epub 2013 Aug 29. PMID 23993888
- [Background] Lloyd-Price J, Abu-Ali G, Huttenhower C. The healthy human microbiome. Genome Med. 2016 Apr 27;8(1):51. doi: 10.1186/s13073-016-0307-y. PMID 27122046